CLINICAL TRIAL: NCT07090616
Title: A Randomized Controlled Trial of the KRONOS Versus Breg T-Scope Post-operative Knee Braces Following Anterior Cruciate Ligament (ACL) Reconstruction
Brief Title: KRONOS Versus Breg T-Scope Post-operative Knee Braces Following Anterior Cruciate Ligament (ACL) Reconstruction
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rush University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 25020201
Record Dates: First submitted 2025-07-21; First posted 2025-07-29 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Anterior Cruciate Ligament (ACL) Reconstruction Surgery
Keywords: Braces; Anterior cruciate ligament (ACL) reconstruction surgery

STUDY DESIGN:
Intervention Model Description: Randomized control trial 1:1 assignment (20 KRONOS Brace: 20 standard of care Breg T-Scope Brace)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Arm 1-Kronos brace (Experimental): Subjects randomized to the treatment group will be measured and fitted with the KRONOS knee brace at their initial clinic visit after study enrollment.
  Interventions: Device: Arm 1-Kronos brace
- Arm 2-Breg T-Scope brace (Active Comparator): Subjects randomized to the standard postoperative Breg T-Scope hinged knee brace in the operating room that will be locked in full extension.
  Interventions: Device: Arm 2-Breg T-Scope brace

INTERVENTIONS:
Device: Arm 1-Kronos brace — Subjects randomized to the treatment group will be measured and fitted with the KRONOS knee brace at their initial clinic visit after study enrollment
  Arms: Arm 1-Kronos brace
Device: Arm 2-Breg T-Scope brace — Subjects randomized to Breg T-Scope Postoperative Brace will be placed in this standard postoperative hinged knee brace in the operating room that will be locked in full extension.
  Arms: Arm 2-Breg T-Scope brace

SUMMARY:
The purpose of this study is to evaluate how well the KRONOS postoperative knee brace reduces pain and enhances recovery compared with the standard Breg T-scope hinged brace following anterior cruciate ligament (ACL) reconstruction knee surgery.

DETAILED DESCRIPTION:
The KRONOS postoperative unloader brace features a new bracing technology that combines the capability of hyperextension immobilization with additional benefits of offloading up to 60 lbs off the knee joint. The adjustable tensioning system in the KRONOS brace offers promising potential to significantly alleviate patient discomfort and pain, facilitate quicker return to a higher level of activity, and ultimately contribute to improved surgical outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Subjects > 18 years of age
* English-speaking
* Scheduled to undergo primary anterior cruciate ligament reconstruction surgery
* No history of prior knee surgery on the operative knee
* No concomitant ligamentous repair or reconstruction procedures (i.e. ligamentous pathology aside from anterior cruciate ligament).
* Subjects undergoing concurrent partial meniscectomy or meniscus repair that would not alter postoperative weight-bearing status or rehabilitation protocol would be eligible for inclusion.
* Clinical and radiographic examination (MRI) consistent with an acute full thickness ACL tear

Exclusion Criteria:

* Age < 18 years of age
* Non-English speaking
* Revision ACL reconstruction
* Multi-ligamentous injury, including concomitant posterior cruciate ligament, medial collateral ligament and fibular collateral ligament injuries
* Concomitant meniscal or cartilage injury that would alter postoperative weight bearing status or rehabilitation protocol
* Inability to comply with the proposed follow-up clinic visits
* Subjects lacking decisional capacity
* Worker's compensation subjects
* Requiring a custom-sized brace

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-02-11 (Actual); Primary Completion 2027-09 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
Rates of extension deficit | 1 year post-operative
  Rates of extension deficit (as measured by the fraction of patients with reduced extension compared to the contralateral determined by heel height and goniometric measurements of knee extension (cm/ degrees)

CONTACTS AND LOCATIONS:
Overall Officials: Jorge Chahla, MD PhD, Principal Investigator — Rush University Medical Center
Locations (1):
- Rush University Medical Center, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No
There is not a plan at this time to make IPD available

DOCUMENTS (1):
  • Study Protocol (2025-04-29): https://cdn.clinicaltrials.gov/large-docs/16/NCT07090616/Prot_000.pdf